CLINICAL TRIAL: NCT06629753
Title: Pilot Implementation of Differentiated Service Delivery for Pregnant and Postpartum Women Living With HIV and Their Infants
Brief Title: Differentiated Service Delivery for Pregnant and Postpartum Women Living With HIV and Their Infants
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, John Moore Humphrey, Assistant Professor of Medicine, Indiana University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 23897; K23HD105495 (NIH)
Record Dates: First submitted 2024-10-02; First posted 2024-10-08 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Hiv; Transmission Vertical; Viremia; Health Care Acceptability; Health Care Utilization
Keywords: prevention of mother-to-child transmission; retention; service delivery; maternal-child health; Kenya
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Viremia; Patient Acceptance of Health Care

STUDY DESIGN:
Intervention Model Description: PPHIV and their children identified who are clinically stable will be differentiated to a care pathway that provides simplified PMTCT services that are adapted to their needs and preferences. PPHIV and their children who are clinically unstable will be differentiated to a care pathway that provides intensified PMTCT services.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DSD arm for stable clients (Experimental): PPHIV who meet the following criteria will be considered stable clients: on current antiretroviral therapy ≥6 months; no active illness in the past 6 months; retained in care; viral load <50 copies/mL within the last 6 months; age ≥18 years; not primigravida; not high-risk pregnancy. PPHIV meeting these criteria will be offered postnatal clinic visits monthly for the first 6 months followed by visits every 2-3 months, flexible ART refills, and encounters with a clinician at each visit and mentor mother as needed. Clients who do not meet these criteria will continue to receive standard-of-care services which include monthly visits and ART refills during pregnancy through 18 months postpartum.
  Interventions: Behavioral: Differentiated service delivery model

INTERVENTIONS:
Behavioral: Differentiated service delivery model — The differentiated service delivery (DSD) intervention is a clinic-level intervention in which PMTCT clients are differentiated into those who are clinically stable or unstable, with each group offered a different package of services to meet their needs. The DSD model that is being tested in this study is an individual-focused, facility-based model designed for implementation within maternal-child health clinics offering integrated HIV services.

SUMMARY:
Differentiated service delivery (DSD) is an evidence-based HIV care and treatment model endorsed by the World Health Organization (WHO) that simplifies HIV services for clients who are clinically stable, improving the quality and efficiency of HIV services. The goal of this implementation-effectiveness pilot study is to evaluate the implementation of a DSD model for pregnant and postpartum women living with HIV and their infants enrolled in care at Huruma Sub-District Hospital in Kenya.

DETAILED DESCRIPTION:
For pregnant and postpartum women living with HIV (PPHIV) in resource-limited settings, maintaining retention in care and viral suppression, and preventing mother-to-child transmission of HIV, are major implementation challenges in the PMTCT cascade. The goal of this study is to execute and evaluate the implementation of a differentiated service delivery (DSD) model for PMTCT to address these challenges. Specifically, this is a pilot study that will evaluate the implementation of a DSD model for PMTCT in a resource-constrained setting in Kenya. The objective of the DSD model is to improve retention in care and viral suppression for PPHIV. In the DSD approach, clinical services are simplified and adapted to the needs and preferences of clients who are clinically stable, allowing the health system to provide intensified services to the clients who unstable according to their needs. Set clinical criteria will be used to determine which PPHIV and their HIV-exposed children are clinically stable and which are unstable. The DSD model will be implemented at Huruma Sub-District Hospital in western Kenya which offers integrated PMTCT services. Over a period of 12 months, all PPHIV that attend this clinic will be recruited to participate in the DSD model as part of the study. The clinical staff will be responsible for triaging PPHIV and their children as stable or unstable according to the DSD eligibility criteria. The implementation success of the DSD model will be determined using the RE-AIM implementation outcomes. This will involve semi-structured interviews with PPHIV and focus group discussions with PMTCT providers participating in the model. Time-motion analysis and medical record review will also be performed to better understand the implementation process and data needed in preparation a future implementation-effectiveness clinical trial. Commensurate with the scope of this pilot implementation study, participants will not be randomized and there will not be a required minimum sample size. The findings from this study will serve as a foundation for a future, large-scale trial to test the effectiveness and implementation of the DSD model for PMTCT in a resource-limited setting.

ELIGIBILITY:
Eligibility criteria for providers:

Inclusion Criteria:

1. ≥18 years of age
2. Able to understand English or Kiswahili
3. Works as a clinician, nurse, peer counsellor, social worker, pharmacist, or clinic supervisor involved in providing PMTCT services in the maternal-child health clinic at Huruma Sub-District Hospital

Exclusion Criteria:

none

Eligibility criteria for PPHIV and their infants enrolled prospectively (n=500)*

Inclusion Criteria:

5. Woman is ≥15 years of age 6. Woman is enrolled in maternal-child health services at HSDH 7. Woman is living with HIV 8. Woman is able to understand English or Kiswahili

Exclusion Criteria:

Cognitive impairment that would impair participation in the study

*All infants born to enrolled women during the study will be included.

Min Age: 1 Day | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 278 (Actual)
Dates: Start 2024-09-13 (Actual); Primary Completion 2025-11-04 (Estimated); Study Completion 2025-11-04 (Estimated)

PRIMARY OUTCOMES:
Number of barriers and facilitators to DSD implementation | One month before implementation of the DSD model in the clinic
  The primary outcome for the analysis in Aim 1 (i.e., the pre-implementation phase) of this study will be the number of barriers/facilitators to implementation as elicited through rapid qualitative analysis of the pre-implementation workshop transcripts
Median difference in number of minutes of PMTCT appointment duration before versus after DSD implementation | One month before and 6 months after implementation of the DSD model in the clinic
  The outcome of interest in this analysis will be the difference in clinic encounter durations (i.e., encounters with clinicians, mentor mother) between clients who are classified as stable versus unstable according to the DSD eligibility criteria, as measured through direct observation and time-motion analysis before an after DSD implementation
Reach | One month before and 6 months after implementation of the DSD model in the clinic
  The proportion of eligible WLH who sign consent to participate in the study among the total number of WLH who attend the PMTCT clinic during the recruitment periods.
Effectiveness, clinic operations level | One month before and during the 12-month period of DSD implementation in the clinic
  The primary outcome will be a ≥20% median reduction in the total clinic visit duration for stable clients compared to their pre-implementation baseline.
Proportion of participants who are virally suppressed <50 copies/mL | One month before and during the 12-month period of DSD implementation in the clinic
  Maternal viral suppression will be assessed among all WLH after enrollment in the study during pregnancy and from delivery to 6 months postpartum, 7-12, and 13-18 months postpartum.
Proportion of children alive and HIV negative | One month before and during the 12-month period of DSD implementation in the clinic
  HIV-free child survival will be assessed among all children of enrolled WLH from birth to 6, 7-12, and 13-18 months postpartum.
Proportion of participants retained in care | One month before and during the 12-month period of DSD implementation in the clinic
  Retention in care will be assessed among all WLH after enrollment in the study during pregnancy and from delivery to 6 months postpartum, 7-12, and 13-18 months postpartum.
Proportion of healthcare workers who adopt the DSD model | During the 12-month period of DSD implementation in the clinic
  The degree to which the clinic commits to and takes on the DSDp model, determined through rapid qualitative analysis of audit/feedback workshop transcripts conducted during the implementation phase
Proportion of PMTCT clients triaged correctly according to the DSD model | During the initial 6 months of DSD implementation in the clinic
  The proportion of PMTCT clients triaged correctly according to the DSD model eligibility criteria.
Proportion of providers affirming the feasibility of the DSD model | During the 12-month period of DSD implementation in the clinic
  The practicality and ease of implementing the DSD model, determined through rapid qualitative analysis of audit/feedback workshop transcripts conducted during the implementation phase
Proportion of providers who perceive the DSD model to be acceptable | During the 12-month period of DSD implementation in the clinic
  How satisfactory or agreeable the DSD model is perceived by its end-users, assessed through structured questionnaires administered to patients and providers.
Proportion of PMTCT clients triaged correctly according to the DSD model at 12 months | At 12 months following the start of DSD implementation in the clinic
  The extent to which a program is part of routine organizational practice, measured through a final time motion analysis and chart review among enrolled participants, conducted over 10 consecutive working days at 6 months at the end of the implementation phase at 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Huruma Sub-District Hospital, Eldoret, Uasin Gishu County, Kenya

IPD SHARING:
Plan to Share IPD: No